CLINICAL TRIAL: NCT06984562
Title: Adaptive Radiation for Locally Advanced Unresectable Pancreatic Cancer: Phase I Dose Escalation Study
Brief Title: Adaptive Radiation for Locally Advanced Unresectable Pancreatic Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RT-221; 25-1011 (Other: FCCC IRB)
Record Dates: First submitted 2025-05-13; First posted 2025-05-22 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-09

CONDITIONS: Locally Advanced Pancreatic Ductal Adenocarcinoma (PDA)
Keywords: Adaptive Radiation Therapy; Pancreatic Ductal Adenocarcinoma; Locally advanced unresectable PDA

STUDY DESIGN:
Intervention Model Description: Adaptive Radiation Therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-Arm (Experimental): Adaptive Radiation Therapy
  Interventions: Radiation: Adaptive Radiation Therapy

INTERVENTIONS:
Radiation: Adaptive Radiation Therapy — Adaptive Radiation Therapy (ART) creates a personalized radiation plan for each treatment session. This means the plan can change from day to day to more precisely target the tumor while protecting the surrounding healthy tissue.
  By closely shaping the radiation to match the tumor's location, ART may reduce the amount of radiation reaching nearby normal tissues. This can allow for higher, more focused doses of radiation to the tumor itself, which may help improve treatment effectiveness while reducing side effects.

SUMMARY:
The goal of this clinical trial is to learn if Adaptive Radiation Therapy (ART) is safe and effective in treating patients with locally advanced pancreatic cancer.

The main questions the study aims to answer are:

* Can ART improve how well radiation therapy targets the most aggressive cancer cells, while protecting the healthy tissue around the tumor?
* Can ART help reduce the side effects that participants may experience during treatment?

Participants will:

* Undergo CT scans to plan the exact location of the radiation treatment. During this process, 1-3 small markers may be placed in or near the tumor to help with the planning.
* Have a tumor biopsy, which involves taking a small sample of tissue from the cancer.
* Receive 5 radiation treatments every other day over a 2-week period.
* Provide blood samples before, during, and after your radiation treatment.

ELIGIBILITY:
Inclusion Criteria

1. Patients must have histologically or cytologically-confirmed PDA.
2. Patients must have locally advanced unresectable PDA.

   • This includes the following- per NCCN criteria*: 2.1 Unreconstructible involvement with the superior mesenteric vein or portal vein due to tumor or bland thrombus OR 2.2 Solid tumor contact with greater than 180 degrees of the superior mesenteric artery or celiac artery OR 2.3. Solid tumor contact with the aorta OR 2.4. Patients with non-metastatic disease that is inoperable by virtue of the operation posing excessive risk to the patient

   *All patients must have been reviewed in the multidisciplinary conference and determined to have unresectable disease by a pancreatic surgeon and to have received or be ineligible for induction chemotherapy based on medical oncology assessment. Documentation of this review in EPIC meeting minutes will satisfy this requirement.
3. Patients enrolled onto the dose escalation arm may have started chemotherapy prior to initiation of radiation therapy and the last dose of chemotherapy must occur at least 2 weeks before start of ART.
4. Eastern Cooperative Oncology Group, or ECOG, performance status 0-2.
5. Adequate bone marrow, hepatic, renal function:

   * ANC ≥ 1,500/µl and PLT ≥ 100,000/µl
   * Bilirubin less than 1.5 ULN
   * AST and ALT < 3X ULN
   * Serum Creatinine <1.5X ULN
6. Women of childbearing potential must not be pregnant (negative pregnancy test within 72 hours prior to registration). Postmenopausal woman must have been amenorrheal and non-lactating for at least 12 months to be considered of non-childbearing potential. Men and women of childbearing potential must be willing to exercise an effective form of birth control (abstinence/contraception) while on study and for at least 6 months after therapy is completed.
7. Age ≥ 18 years
8. Participants must sign a written informed consent and HIPAA consent prior to performance of study-specific procedures or assessments and must be willing to comply with treatment, tissue sample collections, and follow-up.

Exclusion Criteria

1. Radiologically or cytologically confirmed metastatic disease.
2. Patients who have had any prior radiation therapy for pancreatic cancer.
3. Patients who have had prior chemoradiation to an overlapping volume.
4. Patients with adenosquamous carcinoma of the pancreas.
5. Subjects who have had chemotherapy within 2 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 2 weeks earlier to < Grade 2. Patients who received previous immunotherapy or other antibody therapy, within 28 days (immune related toxicities must have resolved to <= Grade 2 prior to starting treatment). Study treatment may be started within these washout periods or with continuing toxicities if considered by the Sponsor-Investigator to be safe and within the best interest of the patient.
6. Concurrent non-study chemotherapy or biologic therapy.
7. A history of ataxia telangiectasia or other documented history of radiation hypersensitivity.

   • Includes both bi- and mono-allelic likely pathogenic or pathogenic ATM mutations (VUS is acceptable).
8. Serious, active infections requiring treatment with IV antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
The rate of acute and late grade ≥3 gastrointestinal toxicity occurring within 3 months of treatment possibly, probably or definitely related to radiation. | From start of radiation to 3 months after the end of radiation treatment

SECONDARY OUTCOMES:
The proportion of patients experiencing local control defined as stable disease or any response at the radiation target site(s). | From the start of radiation to 5 years after end of radiation treatment
Overall Survival Rate - defined as the time from the start of radiation to death or last contact. Individuals who are alive at last follow-up will be considered censored at the time of last contact. | From the start of radiation to death or last contact (up to 5 years after end of treatment).
The rate of acute and late adverse events at time points prescribed in the study calendar using CTCAE version 5.0. | From start of radiation to end of long-term follow up (up to 5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Meyer, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States